CLINICAL TRIAL: NCT07334067
Title: The Application and Efficacy of Dental Prosthesis Membrane in the Preservation of Anterior Esthetic Area After Tooth Extraction
Brief Title: Site Preservation Was Performed Through an Open Healing Oral Restorative Membrane
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Dental Hospital of Zhejiang University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2024-093（R）
Record Dates: First submitted 2025-12-30; First posted 2026-01-12 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2025-12

CONDITIONS: Site Preservation; Soft Tissue Healing; Anterior Dental Aesthetic Area

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control group (Active Comparator): Tooth extraction in the aesthetic area of the anterior teeth with the expansion and flap were reduced in the operative area. Site preservation surgery was performed using Bio-oss (0.5g, Small granule) and bio-gide (25*25mm size) . The gums were closely drawn and sutured.
  Interventions: Procedure: site preservation surgery with close sutures
- Experimental group (Experimental): Tooth extraction in the aesthetic area of the anterior teeth without the expansion and flap were reduced in the operative area. Site preservation surgery was perfomed using Bio-oss (0.5g, Small granule) and Yinlife PCL membrane (25*25mm size) , with opened wound.
  Interventions: Procedure: site preservation surgery with open healing

INTERVENTIONS:
Procedure: site preservation surgery with open healing — Tooth extraction in the aesthetic area of the anterior teeth without the expansion and flap were reduced in the operative area. Site preservation surgery was perfomed using Bio-oss (0.5g, Small granule) and Yinlife PCL membrane (25*25mm size) , with opened wound.
  Arms: Experimental group
Procedure: site preservation surgery with close sutures — Tooth extraction in the aesthetic area of the anterior teeth with the expansion and flap were reduced in the operative area. Site preservation surgery was performed using Bio-oss (0.5g, Small granule) and bio-gide (25*25mm size) . The gums were closely drawn and sutured.
  Arms: Control group

SUMMARY:
In this study, an open healing oral restoration membrane was used for site preservation in the esthetic area after tooth extraction to maintain the space for tooth extraction and bone formation. Clinical observation and cone-beam computed tomography (CBCT) were used to comprehensively evaluate the effect of this operation on promoting the growth of soft and hard tissues, and to provide a new treatment method for site preservation in the esthetic area of clinical anterior teeth.

DETAILED DESCRIPTION:
The anterior tooth region is the key area of aesthetics, which has always been the difficulty and hotspot of implant restoration. In tooth extraction caused by various diseases, the amount of new bone in the tooth extraction fossa often cannot reach the level of the original alveolar ridge, especially the damage to the lip and buccal bone plate is more serious, resulting in insufficient bone mass when the implant is implanted in the later stage. Therefore, bone increment surgery is often used to reconstruct the collapsed alveolar ridge. Among them, site preservation has been widely adopted because of its effective promotion of autologous bone regeneration, simple operation and strong operability. Site preservation is performed by bone grafting on the extraction fossa immediately after tooth extraction to preserve the height and width of the remaining alveolar ridge as much as possible, and retain the corresponding amount of soft tissue, so as to provide sufficient bone mass for later implantation surgery and repair, so as to obtain good aesthetic repair effects.

However, there is currently a lack of oral biofilm that can be opened for healing. After filling bone meal and covering barrier biofilm, the mucosal tissue needs to be fully reduced and then tightly sutured. Sufficient reduction of gingival soft tissue in the aesthetic area of the anterior teeth will undoubtedly increase the surgical wound, and obvious scars will appear in the early stage of repair, seriously affecting the aesthetic appearance. Therefore, in order to simplify the surgical plan of site preservation, reduce trauma, and obtain stable bone growth and good soft tissue morphology, this project proposed to use oral repair membrane with open healing to replace the commonly used clinical collagen membrane for site preservation of the aesthetic area of the anterior teeth.

In this study, an open healing oral restoration membrane was used for site preservation in the esthetic area after tooth extraction to maintain the space for tooth extraction and bone formation. Clinical observation and cone-beam computed tomography (CBCT) were used to comprehensively evaluate the effect of this operation on promoting the growth of soft and hard tissues, and to provide a new treatment method for site preservation in the esthetic area of clinical anterior teeth.

ELIGIBILITY:
Inclusion Criteria:

* 1: Age ≥18 years old

  2: The affected teeth did not have the conditions for immediate implant placement: thin gingival biotype, labial bone plate thickness <1 mm, the labial bone plate was missing, the distance between the labial bone plate crest and the cemento-enamel junction>3 mm

  3: No systemic diseases and good oral hygiene

  4: Be willing to receive treatment and regular follow-up and review, and signed the informed consent

Exclusion Criteria:

* 1: Uncontrolled systemic diseases, such as heart, liver and kidney diseases, systemic infections, diabetes, etc

  2: Women who are pregnant or lactating

  3: Taking bisphosphonates, glucocorticoids and other drugs that affect bone metabolism for a long time or within 5 years

  4: Patients receiving oral and maxillofacial radiotherapy in the past five years

  5: Patients suffering uncontrolled periodontal disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-12-15 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
soft tissue healing efficiency | Immediately after surgery, 7 days, 14 days and 1 month after surgery
  After calibrating the magnification ratio of the tooth extraction wound photos, the reduction ratio of the tooth extraction wound area at 7 days, 14 days, 1 month, and 3 months after surgery was calculated based on the immediate postoperative tooth extraction wound photos to evaluate the soft tissue healing efficiency.

SECONDARY OUTCOMES:
Bone healing efficiency | Preoperative and postoperative 3 months
  NNT Viewer software was used to calibrate CBCT images before and 3 months after surgery. The same section position was used to extract anterior teeth. The area marked by periodontal ligament outside the root before surgery was used as the extraction socket area, and the black corresponding to the blank in the postoperative image was used to represent the unhealed extraction socket. It was used to evaluate the healing efficiency of bone tissue.

CONTACTS AND LOCATIONS:
Locations (1):
- Stomatology Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang, China